CLINICAL TRIAL: NCT05116566
Title: Revealing Information Genuinely & Honestly Across Time: Pediatric Oncology Stakeholder Preferences and Recommendations for Prognostic Communication
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RIGHTime; NCI-2021-12350 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Pediatric Cancer; Communication
Keywords: Prognostic Communication; Advanced Pediatric Cancer; Bereavement; Caregiver; Children; Oncologist; Parents; Young Adults
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients: Three distinct sub-cohorts will be targeted for recruitment to represent perspectives across the advancing illness course: patients ≤3 months from a poor- prognosis diagnosis (cohort 1), patients ≤ 3 months from disease relapse or progression (cohort 2), and patients actively enrolled on a phase I/II trials (cohort 3).For cohorts 1-3, patient-parent dyads will be enrolled when eligible; however, an independent patient is eligible for enrollment if the parent consents for the patient's enrollment but declines his/her own enrollment.
- Parents: Four distinct sub-cohorts of parents will be targeted for recruitment, including cohorts 1-3 and a fourth bereavement cohort. For cohorts 1-3, patient-parent dyads will be enrolled when eligible; however, an independent parent is eligible for enrollment if the patient declines enrollment, but the parent wishes to participate.
- Oncologist: Pediatric oncologists who treat or refer patients for treatment at St. Jude Children's Research Hospital (SJCRH) will be eligible to participate.

SUMMARY:
This study is being conducted to better understand the preferences and recommendations of patients and parents regarding optimal ways to share prognostic communication. Specifically, to learn what stakeholders (i.e., patients, parents, and doctors) believe to be the "right" content, timing, and delivery of this important information.

Specific Aim 1

* To define key stakeholder preferences and recommendations for timing, content, and delivery of prognostic communication across the advancing illness course and bereavement.

Specific Aim 2

* To engage stakeholders in the design of a patient/parent centered RIGHTime framework and communication intervention to promote individualized, timely prognostic disclosure.

DETAILED DESCRIPTION:
This study will have two phases.

Phase 1:

Investigators will define key stakeholder preferences and recommendations for timing, content, and delivery of prognostic communication across the advancing illness course and bereavement. Eligible parents and patients will participate in semi-structured interviews on prognostic communication preferences, stratified by cohort: poor-prognosis diagnosis, advancing disease, phase I/II trial enrollment, and bereavement; eligible oncologists will complete interviews on prognostic disclosure preferences. Participants will participate in a single interview that will last anywhere from 30 to 60 minutes.The interview will be audio-recorded and transcribed. Participant demographic and social determinants of health information will be collected.

Phase 2:

Investigators will partner with a smaller group of stakeholders (parents, patients, and oncologist) from phase 1 to develop a clinical communication guide to help improve communication between patients, families, and cancer doctors. The panel will meet across 4 sessions to develop a conceptual framework that explains the interconnecting variables influencing stakeholder preferences and to design a prognostic communication intervention (i.e., a RIGHTime communication guide) that encourages oncologists to provide individualized, timely prognostic disclosure.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Aged 12-25 years
* Recent diagnosis (< 3 months) of a poor prognosis cancer with an estimated survival of 50% or less by the primary oncologist (cohort 1) OR recent history of disease relapse/progression within the past 3 months (cohort 2) OR active enrollment on a phase I/II trial (cohort 3).
* English-speaking

Parents

* Aged 18 years or older
* Parent (or legal caregiver) of a child with cancer of any age who meets the above criteria for cohorts 1-3 OR of a child who died from cancer 6-24 months from enrollment (cohort 4).
* English-speaking

Oncologists

* Pediatric oncologists who treat patients at SJCRH or who refer patients for treatment to SJCRH

Exclusion Criteria:

* Does not meet the inclusion criteria.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients, parents and Oncologist meeting the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2022-06-18 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Prognostic Communication Preferences | Within 60 days of enrollment
  We will use the rapid analysis (RA) qualitative approach for analysis of interview transcripts methods to define patient, parent, and oncologist preferences and recommendations with respect to timing, content, and delivery of prognostic communication at varying timepoints across the advancing illness course.
Variables influencing stakeholder preferences | After completion of all interviews; 4 sessions over a period of approximately 1-2 years
  We will use a participatory design approach with user-centered design methods, we will convene a Stakeholder Panel comprising patients, parents, oncologists, and researchers that will meet across 4 sessions to develop a conceptual framework that explains the interconnecting variables influencing stakeholder preferences and to design a prognostic communication intervention (i.e., a RIGHTime communication guide) that encourages oncologists to provide individualized, timely prognostic disclosure.

CONTACTS AND LOCATIONS:
Overall Officials: Erica C. Kaye, MD, MPH, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols